CLINICAL TRIAL: NCT07311200
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of D-2570 in Patients With Active Systemic Lupus Erythematosus
Brief Title: A Study of D-2570 in Patients With Active Systemic Lupus Erythematosus (SLE)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2570-205
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Active Systemic Lupus Erythematosus
Keywords: Active Systemic Lupus Erythematosus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: D-2570 and placebo (Experimental)
  Interventions: Drug: D-2570; Drug: D-2570 Placebo
- Group B: D-2570 and placebo (Experimental)
  Interventions: Drug: D-2570; Drug: D-2570 Placebo
- Group C: D-2570 (Experimental)
  Interventions: Drug: D-2570
- Placebo Control Group (Placebo Comparator)
  Interventions: Drug: D-2570 Placebo

INTERVENTIONS:
Drug: D-2570 — Participants will be assigned to one of the following groups: Group A, Group B, Group C, or the placebo control group.
  Arms: Group A: D-2570 and placebo; Group B: D-2570 and placebo; Group C: D-2570
Drug: D-2570 Placebo — D-2570 Placebo
  Arms: Group A: D-2570 and placebo; Group B: D-2570 and placebo; Placebo Control Group

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled Phase II clinical trial designed to evaluate the efficacy and safety of D-2570 in the treatment of active systemic lupus erythematosus.

DETAILED DESCRIPTION:
Subjects who sign the informed consent form will enter the screening period, during which their eligibility will be assessed according to the inclusion and exclusion criteria. Eligible participants who meet the inclusion criteria and do not meet any exclusion criteria will be randomized. Participants will then be assigned to one of the following groups: Group A, Group B, Group C, or the placebo group. They will proceed to the treatment period, during which they will take the corresponding investigational product once daily for 48 consecutive weeks. After completing the treatment, subjects will undergo safety follow-up. Throughout the treatment period, both investigators and subjects will remain blinded. During the study, participants will be required to provide pharmacokinetic and pharmacodynamic blood samples at the time points specified in the trial protocol.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily participates in this study after full informed consent.
* The age is 18 years ≤ age ≤ 70 years, regardless of gender.
* Diagnosed with Systemic Lupus Erythematosus (SLE) at least ≥ 24 weeks prior to screening.
* SLEDAI-2K total score ≥ 8.
* On stable treatment for systemic lupus erythematosus at least 4 weeks prior to randomization, and should remain at a stable dose throughout the trial period.

Exclusion Criteria:

* History of infection as defined in the protocol.
* Any of the medical diseases or disorders listed in the protocol.
* Significant, uncontrolled or unstable disease in any organ.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving the Systemic Lupus Erythematosus Responder Index-4 (SRI-4) at Week 32 | Week 32

SECONDARY OUTCOMES:
Proportion of subjects achieving SRI-4 at Weeks 4, 12, 24, and 48 | Weeks 4, 12, 24, and 48
Proportion of subjects achieving Systemic Lupus Erythematosus Responder Index-6 (SRI-6) at Weeks 4, 12, 24, 32, and 48 | Weeks 4, 12, 24, 32, and 48
Improvement rate in the Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) score from baseline at Weeks 4, 12, 24, 32, and 48 | Weeks 4, 12, 24, 32, and 48
Proportion of subjects with a Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score improvement of ≥50% from baseline at Weeks 4, 12, 24, 32, and 48, among those with a baseline CLASI activity score of ≥10 | Weeks 4, 12, 24, 32, and 48
Proportion of subjects with ≥6 active (tender or swollen) joints at baseline who achieve a reduction of ≥50% in active (tender or swollen) joint count from baseline at Weeks 4, 12, 24, 32, and 48 | Weeks 4, 12, 24, 32, and 48
Proportion of subjects achieving the British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) at Weeks 4, 12, 24, 32, and 48 | Weeks 4, 12, 24, 32, and 48
Proportion of subjects achieving Lupus Low Disease Activity State (LLDAS) at Weeks 4, 12, 24, 32, and 48 | Weeks 4, 12, 24, 32, and 48
Proportion of subjects with a prednisone dose of ≤5.0 mg/day or a reduction of ≥25% from baseline dose during Weeks 44-48 | Weeks 44-48
Changes from baseline of anti-double-stranded DNA (dsDNA) antibody | From enrollment to the end of treatment at 48 weeks
blood drug concentration of D-2570 | From enrollment to the end of treatment at 48 weeks
Incidence of adverse events rate based on NCI CTCAE V5.0 | From enrollment to 52 weeks
Changes from baseline of complement (C3) levels | From enrollment to the end of treatment at 48 weeks
Changes from baseline of complement C4 levels | From enrollment to the end of treatment at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng, Principal Investigator — Zeng

IPD SHARING:
Plan to Share IPD: No